CLINICAL TRIAL: NCT06535971
Title: Effects of Individualized Exercise Intervention Combined With Manual Therapy on Musculoskeletal System, Cardiopulmonary Endurance and Quality of Life in Severe Hemophilia Patients With Polyarthropathy
Brief Title: Individualized Exercise Combined With Manual Therapy in Severe Hemophilia Patients With Polyarthropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111296-E; FarEasternMH (Registry Identifier: WJKao)
Record Dates: First submitted 2024-07-29; First posted 2024-08-02 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-05

CONDITIONS: Severe Hemophilia
Keywords: Physiotherapy; Manual therapy; Exercise
MeSH Terms: conditions — Hemophilia A; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physiotherapy group (Other): Individualized physiotherapy intervention based on manual therapy and exercise 1 session per week for 3 months
  Interventions: Other: Manual therapy combined exercise

INTERVENTIONS:
Other: Manual therapy combined exercise — 1. Manual therapy included fascia release, progressive passive stretch, mobilization, etc.(depend on subject's current condition)
  2. Exercise included muscle strengthening, trunk (spine) stabilization exercise. (depend on subject's current condition)

SUMMARY:
The aim of this study is to investigate the effect of individualized physical therapy, combined manual therapy and exercise intervention, for pain perception, range of motion (ROM), muscle strength, joint health, cardiopulmonary endurance and quality of life (QoL) in patients with severe hemophilia A and multiple hemophilic arthropathy.

DETAILED DESCRIPTION:
The main clinical manifestations of hemophilia are muscle and joint bleeding. Recurrent bleeding leads to a degenerative process known as hemophilic arthropathy. Past studies investigated the effect of manual therapy of exercise for individuals with hemophilia and found to enhance muscle strength, balance, fitness and promote quality of life. However, less study has evaluated the safety and effectiveness of manual therapy combined with exercise for individuals with multiple hemophilic arthropathy. Therefore, the aim of this study is to investigate the effect of individualized physical therapy, combined manual therapy and exercise intervention, for pain perception, range of motion (ROM), muscle strength, joint health, cardiopulmonary endurance and quality of life (QoL) in patients with severe hemophilia A and multiple hemophilic arthropathy.

ELIGIBILITY:
Inclusion Criteria:

* over 20 years old and diagnosed with severe hemophilia
* those who receive prophylaxis regularly
* there are more than 2 target joints (hemophilic arthropathy)

Exclusion Criteria:

* unwilling to sign the informed consent
* any neurological disease or specific musculoskeletal condition (such as fracture) one year ago
* more than 3 (excluding 3) joint replacement surgeries (different joints)
* unable to walk due to hemophilia joint disease or any other diseases
* major bleeding events that pose risks or hinder research
* unable to follow instructions due to cognitive impairment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemophilia Joint Health Score (HJHS) | before intervention (baseline), after intervention 6th week and 12th week
  To measure joint health, in the domain of body structure and function (i.e. impairment), of the joints most commonly affected by bleeding in hemophilia: the knees, ankles, and elbows. It provides a total score (higher score is worse; max=124), joint specific scores, and a global gait score.
Visual Analogue Scale (VAS) | before intervention (baseline), after intervention 6th week and 12th week
  To assess the target joint pain in hemophilia. The minimum value is 0, and the maximum value is 10 (higher score is worse).
6 minute walk test | before intervention (baseline), after intervention 6th week and 12th week
  To evaluate cardiopulmonary endurance. The predictive equation for males: 6MWD(m) = 867 - (5.71 age, yrs) + (1.03 height, cm). The predictive equation for females: 6MWD(m) = 525 - (2.86 age, yrs) + (2.71 height, cm) - (6.22BMI).
Hemophilia Activity List (HAL) | before intervention (baseline), after intervention 6th week and 12th week
  To measure the impact of hemophilia on self-perceived functional abilities in adults.Normalized scores for the domains, components, and the full questionnaire can also be obtained. Missing values are controlled for and the possible scores range from 0 to 100, where 0 represents the worst possible functional status and 100 the best possible functional status.
EQ-5D-5L | before intervention (baseline), after intervention 6th week and 12th week
  To measure the quality of life. Each dimension now has five response levels:
  no problems (1), slight problems (2), moderate problems (3), severe problems (4), unable to/extreme problems (5). The minimum value is 55555 and the maximum value is 11111 (higher score is worse).
  EQ VAS：the minimum score is 0, and the maximum score is 100 (higher score is better).

SECONDARY OUTCOMES:
Daily notes | once a week (each intervention) for 3 months
  record each intervention, such as manual therapy and exercise

CONTACTS AND LOCATIONS:
Overall Officials: Wan Jung Kao, bachelor, Principal Investigator — staff
Locations (1):
- Far Eastern Memorial hospital, New Taipei City, Taiwan

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT06535971/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT06535971/ICF_001.pdf